CLINICAL TRIAL: NCT01973465
Title: Fecal Microbiota Therapy for Recurrent Clostridium Difficile Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, John Farrell, John Farrell M.D., OSF Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSF-13-003
Record Dates: First submitted 2013-10-21; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Clostridium Difficile
Keywords: C-Diff; Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal Microbiota Therapy (Experimental)
  Interventions: Biological: Stool

INTERVENTIONS:
Biological: Stool — Implanting fecal matter via colonscope

SUMMARY:
This study was developed in response to the July, 2013 FDA draft guidance regarding FMT for CDI. The weight of the evidence in the literature suggests that FMT is the most effective treatment for ambulatory outpatients affected by recurrent CDI who fail conventional therapy.

The anticipated benefits to research patients enrolled in this study include resolution of chronic diarrhea, return of bowel habits and nutritional status to normal, and resolution of chronic recurrent CDI.

FMT involves the endoscopic instillation of freshly obtained stool with millions of live bacteria into the recipient's colon by endoscopic lavage. With any endoscopic procedure, there is a risk of perforated viscous. This is very rare, but the risk is increased with severe CDI. The risk of acquisition of communicable enteric or blood borne pathogen appears to be negligible.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. The patient has been treated with appropriate antimicrobial therapy for CDI.
3. The patient has documented relapse/recurrence of infection as demonstrated by positive stool culture, or cytotoxin assay, or PCR toxin assay.
4. Since this study does not involve treatments that have potential teratogenicity, and in general avoidance of antimicrobial treatment during pregnancy is advised (metronidazole is pregnancy category C), women of child-bearing age may be included in the study.

Exclusion Criteria:

- Patients will be excluded from study participation if one of the following categories of exclusion criteria applies:

1. Patient is < 18 years of age
2. Patient has an absolute neutrophil count < 750 cells/mm3.

Stool donors must:

1. be > 18 years of age
2. Complete a screening questionnaire:

   a. One-time donors: Table 1 b. Designated, pre-screened donors: Table 2
3. Be tested for communicable blood-borne and enteric pathogens:

   1. One-time donors: Table 3
   2. Designated, pre-screened donors: Table 4

Table 1: Questionnaire to screen one-time stool donors prior to FMT.

You have been identified as a potential stool donor by __________________ , your (spouse/ son/ daughter/ mother/ father/ life partner), who has been referred for fecal transplantation. Prior to performing the transplantation procedure, the OSF/Saint Francis Medical Center Infection Control Committee requires completion of a screening questionnaire by all potential stool donors:

Your name: ___________________________________________ Date: ___/___/ 2013

Your relationship to the patient: ___________________________ YES / NO

1. Have you ever been diagnosed with Clostridium difficile colitis?
2. Are you currently taking antibiotic medications?
3. Have you been prescribed antibiotics in the past six weeks?

IF the potential stool donor answers YES to questions 1, 2, or 3 - please STOP.

Do you have a history of any of the following: (Please Circle)

Hepatitis A YES / NO Hemophilia YES / NO Hemodialysis treatment YES / NO Rejected or refused blood donation YES / NO HIV/AIDS YES / NO Hepatitis B YES / NO Hepatitis C YES / NO Use of intravenous drugs or medications YES / NO Incarceration YES / NO Abnormal blood tests of liver enzymes YES / NO Accepting money or drugs in exchange for sex YES / NO Receipt of a blood transfusion between 1977 - 1992 YES / NO Infectious gastroenteritis or diarrhea YES / NO

Did you answer YES to any of the above? YES / NO

Table 2: Questionnaire to screen designated stool donors prior to each FMT.

You have been identified as a potential stool donor for a patient who has been referred to Saint Francis Medical Center for fecal transplantation. Prior to performing the transplantation procedure, the OSF/Saint Francis Medical Center Infection Control Committee requires completion of a screening questionnaire by all potential stool donors:

Your name: ___________________________________________ Date: ___/___/ 2013

Your relationship to the patient: ___________________________ YES / NO

1. Have you ever been diagnosed with Clostridium difficile colitis?

4. Are you currently taking antibiotic medications?

5. Have you been prescribed antibiotics in the past six weeks?

IF the potential stool donor answers YES to questions 1, 2, or 3 - please STOP.

Do you have a history of any of the following: (Please Circle)

Hepatitis A YES / NO Hemophilia YES / NO Hemodialysis treatment YES / NO Rejected or refused blood donation YES / NO HIV/AIDS YES / NO Hepatitis B YES / NO Hepatitis C YES / NO Use of intravenous drugs or medications YES / NO Incarceration YES / NO Abnormal blood tests of liver enzymes YES / NO Accepting money or drugs in exchange for sex YES / NO Receipt of a blood transfusion between 1977 - 1992 YES / NO Infectious gastroenteritis or diarrhea YES / NO

Did you answer YES to any of the above? YES / NO

Table 3: Required stool donor screening laboratory studies prior to FMT

Stool:

Giardia & Cryptosporidium stool antigen testing Stool ova & parasite testing Cultures for Salmonella, Shigella and E. coli O157:H7 Clostridium difficile toxin B PCR assay

Blood:

HIV 1&2 Ab/Ag HAV IgM Ab HBV core Ab & Ag HCV Ab HTLV-1 Ab

Table 4: Laboratory studies every 120 days for designated stool donors

Stool:

Giardia & Cryptosporidium stool antigen testing Stool ova & parasite testing Cultures for Salmonella, Shigella and E. coli O157:H7 Clostridium difficile toxin B PCR assay

Blood:

HIV 1&2 Ab/Ag HAV IgM Ab HBV core Ab & Ag HCV Ab HTLV-1 Ab

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Weight and Number of bowel movements/day | 30 and 90 days
  In the present study we will record each subjects weight and number of bowel movements/day prior to FMT and following FMT at 30 and 90 days.

SECONDARY OUTCOMES:
Evaluate the most appropriate patient population for FMT | 30 and 90 days
  Our study will include ambulatory outpatients as well as hospitalized, debillitated patients. FMT has demonstrated effectiveness (both systematic reviews and RCT) for treatment of recurrent Clostridium difficile infection in ambulatory outpatient populations. A secondary outcome of our study is to evaluate stratify our patient population and examine FMT success rates for out two primary outcome measures in outpatients vs. inpatients.
Determine the overall success of FMT | 30 and 90 days
  An additional secondary outcome measure will be to examine the percent of patients who undergo 2nd or third FMT. and the success rate (in terms of primary outcome measures) for each subsequent FMT.

CONTACTS AND LOCATIONS:
Overall Officials: John J Farrell, M.D., Principal Investigator — OSF Healthcare System
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

REFERENCES:
- [Background] Hall IC, O'Toole E. Intestinal flora in newborn infants with a description of a new pathogenic anaerobe, Bacillus difficilis. Am J Dis Child 1935;49:390-402.
- [Background] Bartlett JG, Chang TW, Gurwith M, Gorbach SL, Onderdonk AB. Antibiotic-associated pseudomembranous colitis due to toxin-producing clostridia. N Engl J Med. 1978 Mar 9;298(10):531-4. doi: 10.1056/NEJM197803092981003. PMID 625309
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Background] True E, Tsoraides S, Bonello JP. Fecal Microbiota Therapy in the Treatment of Clostridium difficile diarrhea. 63rd Annual Scientific Meeting, Illinois Chapter, American College of Surgeons. June 7, 2013.
- [Background] Sax, PE. NEJM Journal Watch. http://blogs.jwatch.org/hiv-id-observations/index.php/fda-fecal- transplants-need-investigational-new-drug-application/2013/05/12/